CLINICAL TRIAL: NCT03974139
Title: Study of the Communication of the Hypothalamus With the Periphery: Impact of Metformin on Leptin Transport in the Cerebrospinal Fluid of Obese Patients. A Monocentric Prospective Study
Brief Title: Impact of Metformin on Leptin Transport in Cerebrospinal Fluid of Obese Patients
Acronym: LEPTOB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC-P0054
Record Dates: First submitted 2019-05-28; First posted 2019-06-04 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Obesity Without Type 2 Diabetes, With BMI>30
Keywords: metformin; leptin; cerebrospinal fluid
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese patients (Experimental): Patients with body mass index >30
  Interventions: Drug: Metformin Oral Tablet

INTERVENTIONS:
Drug: Metformin Oral Tablet — Day 1 to day 3: 500 mg/day Day 4 to day 6: 500 mg/twice a day Day 7 to day 9: 500 mg three times a day Day 10 until next lumbar puncture : 850 mg three times a day

SUMMARY:
Obesity, a major health problem, is gradually transforming into a global epidemic. The current obesity treatment with long term efficacy is the bariatric surgery, however, the operative risk of this procedure is high and the post-operative iotrogeny may be important. Obesity is most often associated to the feeding behavior which depends on hypothalamic integration of peripheral signals such as leptin and glucose. High levels of circulating leptin are detected in obese patients. These elevated leptin levels fail to reduce appetite or increase energy expenditure. The mechanism underlying this non-integration of peripheral signals remains to be identified. The ratio of leptin levels in the cereprospinal fluid (CSF) and in the periphery is drastically decreased in obese patients when compared to lean individuals, therefore a defective transport of circulating leptin into the brain via the CSF is maybe linked to obesity.

DETAILED DESCRIPTION:
We hypothesize that the alteration of leptin transport into the CSF of obese patients could be modulated by drugs such as metformin which is widely used worldwide to treat diabetes. This study is monocentric, prospective, one-arm type and interventional. The main objective isto evaluate the impact of metformin on the transport of leptin into the CSF of obese patients.

We propose to show a variation of CSF leptin / serum leptin before and after metformin treatment and study its association with changes in hypothalamic metabolic activity, cognitive and appetite-related behaviors and ratio of other metabolic signals. This would support the hypothesis of modulation of resistance to peripheral leptin by metformin and thus uncover a new indication for metformin treatment towards the management of obesity.

For this purpose, volunteers will be subjected to blood sampling via venipuncture, CSF collection via lumbar puncture, MRI assessments and questionnaires (cognitive tests, food survey and feeding behavior) before and after a 3-month metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 40 years old
* Body mass index >30
* For childbearing age women: use of an effective contraceptive method for the duration of the study
* Patients willing to participate in the study and who have signed the informed consent form
* Patients with health insurance

Exclusion Criteria:

* Genetic obesity
* Type 2 diabetes defined by 2 fasting blood glucose >1,26g/L or blood glucose >2 g/L at 120 min of oral glucose tolerance test with 75 g of glucose
* Patients already treated with metformin
* Type 1 diabetes
* Active neoplastic pathology, diagnosed < 5 years, or in treatment
* Neurological pathology (demyelinating, tumor, vascular)
* Adipose tissue pathology (lipodystrophy)
* History of bariatric surgery
* Contraindication to metformin
* Lumbar puncture contraindication
* MRI contraindication
* Person unable to consent, or benefiting from a legal protection regime (guardianship/curatorship/guardianship of justice)
* Pregnant or breastfeeding woman
* Contra-indication to impedance measurement
* Contraindication to indirect calorimetry: claustrophobia
* Taking a psychotropic drug

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
cerebrospinal fluid /plasma leptin ratio | 3 months

SECONDARY OUTCOMES:
cerebrospinal fluid /plasma glucose ratio | at day 0, 3 months
cerebrospinal fluid /plasma glucagon like peptide 1 (GLP1) ratio | at day 0, 3 months
cerebrospinal fluid /plasma insulin ratio | 3 months
cerebrospinal fluid /plasma ghrelin ratio | at day 0, 3 months
Cerebrospinal fluid levels of Agouti-Related Peptide (AgRP) | at day 0, 3 months
Plasma levels of Agouti-Related Peptide (AgRP) | at day 0, 3 months
Cerebrospinal fluid levels of proopiomelanocortin (POMC) | at day 0, 3 months
Plasma levels of proopiomelanocortin (POMC) | at day 0, 3 months
Cerebrospinal fluid levels of neuropeptide Y (NPY) | at day 0, 3 months
Plasma levels of neuropeptide Y (NPY) | at day 0, 3 months
Cerebrospinal fluid levels of leptin soluble receptor | at day 0, 3 months
Plasma levels of leptin soluble receptor | at day 0, 3 months
Apparent diffusion coefficient (ADC) | at day 0, 3 months
  Apparent diffusion coefficient (ADC) is a measure of the magnitude of diffusion (of water molecules) within tissue, and is commonly clinically calculated using Magnetic resonance imaging (MRI). An ADC of a tissue is expressed in units of mm2/s
Hypothalamic concentration of N-acetyl-aspartate (NAA) | at day 0, 3 months
  This concentration will be measure by spectroscopy
Hypothalamic concentration of creatine | at day 0, 3 months
  This concentration will be measure by spectroscopy
Hypothalamic concentration of Choline | 3 months
  This concentration will be measure by spectroscopy
Hypothalamic concentration of Glutamine / glutamate | at day 0, 3 months
  This concentration will be measure by spectroscopy
Hypothalamic concentration of gamma-aminobutyric acid (GABA) | at day 0, 3 months
  This concentration will be measure by spectroscopy
Weight | at day 0, 3 months
Abdominal circumference | 3 months
Percentage of body fat | at day 0, 3 months
  This parameter will measure by bioelectrical impedance analysis (BIA). A weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body.
Fat free mass (Kg) | at day 0, 3 months
  This parameter will measure by bioelectrical impedance analysis (BIA). A weak electric current flows through the body and the voltage is measured in order to calculate impedance (resistance) of the body.
Energy expenditure | at day 0, 3 months
  This parameter will measure by indirect calorimetry (kCal / 24h)
Score of the Three Factor Eating Questionnaire (TFEQ) | 3 months
  The TFEQ contains 51 items and measures three dimensions of eating behavior:
  * cognitive restraint of eating' (Factor I - 21 items)
  * disinhibition (Factor II - 16 items)
  * hunger (Factor III - 14 items)
  Each item scores either 0 or 1 point. The minimum score for factors I-II-III is therefore 0-0-0, the possible maximum score 21-16-14
Score of the Dutch Eating Behaviour Questionnaire (DEBQ) | at day 0, 3 months
  This is a 33-item self-report questionnaire to assess three distinct eating behaviors in adults: (1) emotional eating, (2) external eating, and (3) restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Prévot, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Vincent Florent, MD, MSc, PhD, Principal Investigator — Centre Hospitalier d'Arras, INSERM
Locations (1):
- Centre hospitalier d'Arras, Arras, France

IPD SHARING:
Plan to Share IPD: Undecided